CLINICAL TRIAL: NCT00262288
Title: A Phase II/III Study of the Efficacy and Safety of Recombinant Human C1 Inhibitor for the Treatment of Acute Attacks in Patients With Hereditary Angioedema
Brief Title: Recombinant Human C1 Inhibitor for the Treatment of Acute Attacks in Patients With Hereditary Angioedema
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1 1203-01
Record Dates: First submitted 2005-12-01; First posted 2005-12-06 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Genetic Disorders
MeSH Terms: conditions — Genetic Diseases, Inborn

ARMS (1):
- Recombinant Human C1INH (Experimental)
  Interventions: Drug: i.v. recombinant human C1 inhibitor

INTERVENTIONS:
Drug: i.v. recombinant human C1 inhibitor
  Other Names: rhC1INH

SUMMARY:
The purpose of this multi-center study is to explore the efficacy, safety, tolerability and pharmacokinetics/pharmacodynamics of recombinant human C1 inhibitor in the treatment of acute attacks in patients with hereditary angioedema.

ELIGIBILITY:
Main inclusion Criteria:

* Clinical and laboratory diagnosis of HAE
* Plasma level of functional C1INH of less than 50% of normal
* Severe attack of abdominal, facial-oro-pharyngeal, genito-urinary and/or peripheral HAE.

Main exclusion Criteria:

* Acquired angioedema
* Pregnancy or breastfeeding
* Participation in another clinical study within prior 3 months

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-04; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Primary outcomes: Relief of angioedema symptoms | 24 hours

SECONDARY OUTCOMES:
Secondary outcomes: Safety and tolerability; pharmacokinetics/pharmacodynamics | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jan Nuijens, MD, PhD, Study Chair — Pharming Technologies B.V.
Locations (1):
- For information on sites in Europe, please contact Pharming Technologies., Leiden, Netherlands